CLINICAL TRIAL: NCT06920758
Title: A 6-month, Randomized, Double-blind, Placebo Controlled Study Evaluating the Efficacy and Safety of USPlus DERM to Promote Hair Growth in Men and Women With Self-perceived Thinning Hair.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ablon Skin Institute Research Center (Other)
Collaborators: U.S. Nutraceuticals, Inc. dba Valensa International (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VAL-HT-002
Record Dates: First submitted 2025-04-03; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Thinning Hair
Keywords: Thinning hair, hair loss, hair shedding
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- USPlus DERM softgels (Active Comparator): USPlus® DERM Bioactive Fatty Acids 160 mg Softgels
  Interventions: Dietary Supplement: USPlus DERM Bioactive Fatty Acids 160 mg Softgels
- Placebo softgels (Placebo Comparator): Placebo Softgels
  Interventions: Other: Placebo softgel

INTERVENTIONS:
Dietary Supplement: USPlus DERM Bioactive Fatty Acids 160 mg Softgels — USPlus® DERM Bioactive Fatty Acids (160 mg) Ingredient List (Per Softgel)
  Active: 100% Concentrated Lipidosterolic Extract of Saw Palmetto (Serenoa repens).
  Shell: Bovine Gelatin, Glycerin, Water
  Arms: USPlus DERM softgels
Other: Placebo softgel — Placebo Ingredient List:
  Palm oil Gelatin Glycerin Water Caramel color
  Arms: Placebo softgels

SUMMARY:
The goal of this clinical trial is to substantiate the effectiveness and safety of USPlus® DERM for self-perceived thinning hair compared to placebo in healthy men and women ages 25-65 over the course of six months of continued use. Participants will be asked to have attend three office visits, one phone call, have photos taken of their hair and answer questionnaires related to their thinning hair.

DETAILED DESCRIPTION:
Hair shedding and thinning is presenting at alarming rates. It affects over 80% of men and 50% of women in the United States alone. As a multifactorial condition, while genetics is a small component, change in environmental exposures, nutrition, hormones, stress and lifestyle play significant roles. Currently, many individuals are looking for natural or prescription free options to combat challenges in hair thinning. One of the main ingredients added to current formulations is the natural supplement Saw Palmetto (Serenoa repens). To maintain thick full hair takes work, and prevention of hair thinning, shedding and hair loss requires early intervention. This study is performed to demonstrate the success of a long-standing supplement in the hair loss treatment armamentarium.

Oral medications come with significant side effects, and other modalities like laser and platelet rich plasma can be expensive to afford. Supplements therefore become a great natural alternative. Saw palmetto or Serenoa repens is a plant from the Areaceae family also known as Sabal serrulataa that acts as a competitive nonselective inhibitor of 5-alpha reductase (5αR) types I and II, which blocks the conversion of testosterone to its active metabolite, dihydrotestosterone. This process has been shown to help prevent miniaturization of hairs that lead to hair loss. Valensa International has analyzed the vast amount of science, as well as their own research data, to understand the impact of USPlus® DERM which contains concentrated lipidosterolic extracts of saw palmetto on hair health. The mechanism of action appears to prolong the anagen phase, tends to enhance dermal papilla, and maintains the follicle stem cell niche. USPlus® DERM is concentrated in bioactive free fatty acids (the building blocks of hair) and can help benefit hair health, the hair growth cycle and hair characteristics. Since hair loss has a multifactorial etiology, studying USPlus® DERM in the treatment

The purpose of this clinical research study is to evaluate the efficacy and safety of USPlus® DERM compared to placebo in sixty (60) healthy male and female subjects, 25-65 years of age with self-perceived hair thinning over the course of six (6) months of continued use.

Pre-Study Procedures

1. Candidate subjects will be screened with selected eligibility requirements by telephone prior to Visit 1. The questions include the following: (1) Are you between the ages of 25-65? (2) Do you feel that your hair is thinning? 3) Are you able to attend periodic visits at your study doctor's office (3 visits and one phone call over a 6 month period)?
2. Candidate subjects will be assigned an appointment time for visiting the clinic.

VISIT PROCEDURES

Visit 1: Baseline, Day 0

1. Individuals will be given an informed consent form (ICF) document, HIPAA form and Photography release form to read. They will have all of their study related questions answered by the Investigator and if they agree, they will sign the ICF, HIPAA and Photography release forms. Subjects will be given one copy of the signed ICF, HIPAA and Photography release forms to keep. The original documents will remain at Ablon Skin Institute and Research Center in the subject's file.
2. Investigator and/or Study Coordinator will review with subject and complete the checklist for demographics, medical history and previous/concomitant medications.
3. Investigator and/or Study Coordinator will review with subject and complete the checklist for all inclusion and exclusion criteria.
4. Subjects will receive a brief physical exam, including examination of the scalp, to rule out any immediately observable medical issues and scalp disorders that are unacceptable for qualification in accordance with the study exclusion criteria. The physical will additionally include vital signs (blood pressure, heart rate, respiration rate, and temperature), weight and height. Subjects hair thinning will be rated by the Investigator using either the Norwood Scale for men or the Savin Pictorial Scale for women.
5. Subjects who are female of childbearing potential will have a urine pregnancy test performed.
6. Subjects who have completed all the initial paperwork and meet the inclusion/exclusion qualifications (including findings of the physical exam) will be assigned a unique subject number. Subjects will be randomized to a treatment group.
7. Subjects will have Canfield Intellistudio 2-D digital photography of their entire head/hair region to assess overall general hair growth and fullness.
8. Subjects will have two (2) target sites selected and measured by the Investigator.
9. Subjects will have Canfield HairMetrix trichoscopy imaging of the two (2) target site areas taken for hair analysis.
10. Subjects will have a Hair Shedding Pull test in four regions of the hair by the Investigator.
11. Subjects will complete the Hair Thinning Quality of Life Questionnaire.
12. Subjects will be dispensed a three (3) month supply of the Active or Placebo and given written and verbal Usage and Lifestyle instructions.
13. Subjects will be given their next appointment date and time, and instructed to bring back all Study IP, including empty bottles.

Phone Call: Day 56 ± 2 days

1. The Study Coordinator will ask subjects if they have experienced any changes in their health or taken new/adjusted current medications since the last visit. If an AE or SAE is reported, the examining Investigator will be informed and the appropriate forms will be completed.
2. The subjects will be asked about the amount of unused Study IP that they have in their current bottles to determine subject compliance with the protocol and usage instructions. Subjects found to be consistently out of compliance will be reminded of the correct usage instructions. Non-compliance will be noted in the Subject IP Compliance Log.
3. Subjects will be asked a series of hair self-assessment questions and hair thinning quality of life questions. The answers to the questionnaires will be recorded in the subject file by the Study Coordinator.
4. Subjects will be reminded of their next appointment date and time, and instructed to bring back all Study IP, including empty bottles to their next appointment.

Visit 2: Day 90 (± 7 days)

1. The Study Coordinator will ask subjects if they have experienced any changes in their health or taken new/adjusted current medications since the last visit. If an AE or SAE is reported, the examining Investigator will be informed and the appropriate forms will be completed.
2. The unused Study IP will be collected and counted to determine subject compliance with the protocol and usage instructions. Subjects found to be consistently out of compliance will be reminded of the correct usage instructions. Non-compliance will be noted in the Subject IP Compliance Log.
3. The subject will have their weight, blood pressure, heart rate, respiratory rate and temperature monitored and recorded in the source.
4. Subjects will have Canfield Intellistudio 2-D digital photography of their entire head/hair region to assess overall general hair growth and fullness.
5. Subjects will have Canfield HairMetrix trichoscopy imaging of the two (2) target site areas taken for hair analysis.
6. Subjects will have a Hair Shedding Pull test in four regions of the hair by the Investigator.
7. Subjects will have their hair assessed by the Investigator for Hair Growth and Hair Quality.
8. Subjects will complete the Hair Self-Assessment Questionnaire and the Hair Thinning Quality of Life Questionnaire.
9. Subjects will be dispensed a three (3) month supply of the Active or Placebo and given written and verbal Usage and Lifestyle instructions.
10. Subjects will be given their next appointment date and time, and instructed to bring back all Study IP, including empty bottles.

Visit 3: Day 180 (± 7 days)

1. The Study Coordinator will ask subjects if they have experienced any changes in their health or taken new/adjusted current medications since the last visit. If an AE or SAE is reported, the examining Investigator will be informed and the appropriate forms will be completed.
2. The unused Study IP will be collected and counted to determine subject compliance with the protocol and usage instructions. Non-compliance will be noted in the Subject IP Compliance Log.
3. The subject will have their weight, blood pressure, heart rate, respiratory rate and temperature monitored and recorded in the source.
4. Subjects will have Canfield Intellistudio 2-D digital photography of their entire head/hair region to assess overall general hair growth and fullness.
5. Subjects will have Canfield HairMetrix trichoscopy imaging of the two (2) target site areas taken for hair analysis.
6. Subjects will have a Hair Shedding Pull test in four regions of the hair by the Investigator.
7. Subjects will have their hair assessed by the Investigator for Hair Growth and Hair Quality.
8. Subjects will complete the Hair Self-Assessment Questionnaire, Hair Thinning Quality of Life Questionnaire and the Hair Product Subject Satisfaction Questionnaire.
9. Subjects will be compensated for their participation in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females of all Fitzpatrick Skin Types between 25 and 65 years of age.
2. Subjects must be willing to provide verbal understanding and sign an Informed Consent Form, HIPAA Form and Photography Release Form approved by the Institutional Review Board.
3. Subjects must be in general good health, as determined by the Investigator.
4. Subjects with self-perceived hair thinning as determined on initial study assessment by the Investigator (excluding patients with medically diagnosed telogen effluvium).
5. Subjects willing to undergo a brief physical exam to include height, weight, blood pressure, pulse, physical scalp exam and basic systems evaluation (Skin, Respiratory, Cardiovascular, Gastrointestinal, Endocrine, Neurological and Musculoskeletal systems) by the Investigator.
6. Male subjects with frontal and/or vertex patterns I, II, IIA, III, III vertex and IV during the physical scalp exam by the Investigator rated based on the Norwood Classification Scale.
7. Female subjects with I-1, I-2 and I-3 during the physical scalp exam by the Investigator rated based on the Savin Pictorial Scale.
8. Subjects willing to not substantially change their current diet, medications, dietary supplements and exercise routines for the duration of the study. If a subject receives physician guidance during the study to change diet, medications, supplements or exercise routine, the subject will need to notify the clinic as soon as possible.
9. Females of child bearing potential (FOCBP) must be willing to have a urine pregnancy test and practice effective contraception for the duration of the study. (Effective contraception is defined as stabilized on oral contraceptive for at least 3 months as of the start of the study, intrauterine device, condom with spermicide, diaphragm with spermicide, implant, NuvaRing®, injection, transdermal patch or abstinence.) Females on birth control pills must have taken the same type of pill for at least 3 months prior to entering the study and must not change type during the study. Those who have used birth control pills in the past must have discontinued usage at least 3 months prior to the start of the study. The initiation of birth control should not have been associated with the initiation of hair loss/thinning.
10. FOCBP must have a negative urine pregnancy test at the Baseline Visit.
11. Subjects willing to have 2-D digital photography of the entire head/hair region for overall evaluation of general hair growth and quality by the Investigator.
12. Subjects willing to have digital trichoscopy photography of the target site areas on the scalp for analysis of hair counts and other hair measurements.
13. Subjects must be willing and able to complete and understand the rating questionnaires.
14. Subjects must maintain a consistent length, cut, style and color throughout the six (6) month study period.
15. Subjects who have color treated hair must be willing to have the color treatment performed at the same time interval prior to each visit (i.e. If on Visit 1 the color treatment was done one week prior then the color treatment is expected to occur at a similar interval of one week prior to Visits 2 and 3).
16. Subjects willing to maintain their normal hair shampooing frequency, use a mild non-medicated shampoo and conditioner for the duration of the study and attend visits with clean and dry hair (shampoo must be done 24 hours or more prior to the visit).
17. Subjects must be willing and able to attend all study visits and comply with the study product daily usage and lifestyle instructions.

Exclusion Criteria:

1. Subjects who are pregnant, nursing mothers, planning a pregnancy during the course of the study, or become pregnant during the study.
2. Male subjects with male pattern hair loss with frontal and/or vertex patterns IIIA, IVA, V, VA, VI, VII ratings using the Norwood Classification Scale as determined during the physical scalp exam by the Investigator.
3. Female subjects with I-4, II-1,II-2, III Advanced and Frontal ratings using the Savin Pictorial Scale as determined during the physical scalp exam by the Investigator.
4. Subjects who have had a hair transplant.
5. Subjects with hair extensions or who are planning on getting hair extensions during the duration of the study.
6. Subjects with any known allergy or sensitivity to any shampoo and/or conditioner.
7. Subjects with a known stressful incident within the last six months (e.g. death in family, miscarriage).
8. Subjects who have recently (within the last 3 months) started the use of hormones for birth control or hormone replacement therapy (HRT). Women currently using hormones for birth control or HRT must have been on a stable dose (3 months or longer) in order to be eligible for the study.
9. Subjects using Low Level Laser Therapy (LLLT) or other light therapy to treat thinning hair in the last 3 months.
10. Subjects who have regularly used Rogaine (Minoxidil), Nioxin and /or Finasteride or undergone any other hair or scalp treatments within the last 3 months.
11. Subjects who have used prescription drugs known to affect the hair growth cycle within the last 3 months (e.g., hormone-based birth control for less than 3 months, cyproterone acetate, aldactone/spironolactone or any 5-alpha-reductase inhibitor).
12. Subjects who have regularly used anti-androgenic therapies (i.e. spironolactone, flutamide, cyproterone acetate, progesterone and/or bicalutamide) or undergone any other hair or scalp treatments within the last 3 months.
13. Subjects suffering from other hair loss disorders, such as alopecia areata, scarring alopecia, androgenetic alopecia and telogen effluvium as determined during initial study assessment and physical scalp exam by the Investigator.
14. Subjects with self-reported uncontrolled diseases (i.e. diabetes, hypertension, hyperthyroidism, hypothyroidism, etc.). Whether medical conditions are under control with or without treatment will be assessed on an individual basis by the Investigator based on her medical and clinical expertise.
15. Subjects with self-reported active hepatitis, immune deficiency, HIV or autoimmune disease.
16. Subjects having a known active dermatologic condition of the scalp that may place the subject at a greater risk or interfere with clinical evaluations (ie. seborrheic dermatitis, psoriasis, atopic dermatitis, advanced skin cancer, etc.) as determined by the Investigator based on her medical and clinical expertise.
17. Subjects who are unable to communicate or cooperate with the Investigator due to language problems, poor mental development, or impaired cerebral function.
18. Subjects with any underlying disease that the Investigator deems uncontrolled, and poses a concern for the subject's safety while participating in the study.
19. Subjects with use of any medications that are known to potentially cause hair loss or affect hair growth as determined by the Investigator based on her medical and clinical expertise.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-12-16 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Change in terminal hair counts from Baseline to Day 180 using the Canfield HairMetrix system. | Baseline to Day 180
  Change in terminal hair counts from Baseline to Day 180 using the Canfield HairMetrix system. A statistically significant increase in count at Day 180 in comparison to Baseline for subjects who were assigned to the Active compared to subjects who were assigned to the placebo indicates an improvement for the indicated parameter.
Change in vellus hair counts from Baseline to Day 180 using the Canfield HairMetrix system. | Baseline to Day 180
  Change in vellus hair counts from Baseline to Day 180 using the Canfield HairMetrix system.
Change in total hair counts from Baseline to Day 180 using the Canfield HairMetrix system. | Baseline to Day 180
  Change in total hair counts from Baseline to Day 180 using the Canfield HairMetrix system. A statistically significant increase in count at Day 180 in comparison to Baseline for subjects who were assigned to the Active compared to subjects who were assigned to the placebo indicates an improvement for the indicated parameter.

SECONDARY OUTCOMES:
Change in terminal to vellus ratio using the Canfield HairMetrix system from Baseline to Day 180. | Baseline to Day 180
  A statistically significant increase in terminal to vellus ratio at Day 180 in comparison to Baseline for subjects who were assigned to Active compared to subjects who were assigned to the placebo indicates an improvement for the indicated parameter.
Change in average hairs per follicular unit using the Canfield HairMetrix system from Baseline to Day 180. | Baseline to Day 180
  A statistically significant increase in average hairs per follicular unit at Day 180 in comparison to Baseline for subjects who were assigned to Active compared to subjects who were assigned to the placebo indicates an improvement for the indicated parameters.
Change in average hair width (μm) using the Canfield HairMetrix system from Baseline to Day 180. | Baseline to Day 180
  A statistically significant increase in score of average hair width (μm) at Day 180 in comparison to Baseline for subjects who were assigned to Active compared to subjects who were assigned to the placebo indicates an improvement for the indicated parameters.
Change in follicular units per cm² using the Canfield HairMetrix system from Baseline to Day 180. | Baseline to Day 180
  A statistically significant increase in score of follicular units per cm² at Day 180 in comparison to Baseline for subjects who were assigned to Active compared to subjects who were assigned to the placebo indicates an improvement for the indicated parameters.
Change in inter-follicular mean distance (mm) using the Canfield HairMetrix system from Baseline to Day 180. | Baseline to Day 180
  A statistically significant decrease in score of inter-follicular mean distance (mm) at Day 180 in comparison to Baseline for subjects who were assigned to Active compared to subjects who were assigned to the placebo indicates an improvement for the indicated parameter.
Investigator Hair Quality Global Improvement Scale | Baseline to Day 180
  Investigator Hair Quality Global Improvement Scale scores assessed by Investigator using Canfield Intellistudio standardized 2D photographs to assess changes from Baseline to Day 180. A positive score at Day 180 for subjects who were assigned to the Active compared to subjects who were assigned to the placebo indicates an improvement for the indicated parameters.
Investigator Hair Growth Global Improvement Scale | Baseline to Day 180
  Investigator Hair Growth Global Improvement Scale scores assessed by Investigator using Canfield Intellistudio standardized 2D photographs to assess changes from Baseline to Day 180. A positive score at Day 180 for subjects who were assigned to the Active compared to subjects who were assigned to the placebo indicates an improvement for the indicated parameters.
Change in Hair Shedding Pull Test scores | Baseline to Day 180
  Change in Hair Shedding Pull Test scores from Baseline to Day 180. A statistically significant decrease in count at Day 180 in comparison to Baseline for subjects for subjects who were assigned to the Active compared to subjects who were assigned to the placebo indicates an improvement for the indicated parameter.
Improvement in Hair Self-Assessment Questionnaire | Baseline to Day 180
  Improvement in Hair Self-Assessment Questionnaire from Baseline to Day 180. A statistically significant increase in score at Day 180 in comparison to Baseline for subjects who were assigned to the Active compared to subjects who were assigned to the placebo indicates an improvement for the indicated parameter.
Improvement in Hair Thinning Quality of Life Questionnaire | Baseline to Day 180
  Improvement in Hair Thinning Quality of Life Questionnaire from Baseline to Day 180. A statistically significant decrease in score at Day 180 in comparison to Baseline for subjects who were assigned to the Active compared to subjects who were assigned to the placebo indicates an improvement for the indicated parameter.
Favorable Analysis of the Hair Product Subject Satisfaction Questionnaire | Baseline to Day 180
  at Day 180. Favorable analysis at Day 180 for subjects who were assigned to the Active compared to subjects who were assigned to the placebo would be indicated by high response values.

CONTACTS AND LOCATIONS:
Overall Officials: Glynis Ablon, MD, FAAD, PI, Principal Investigator — Ablon Skin Institute Research Center
Locations (1):
- Ablon Skin Institute and Research Center, Manhattan Beach, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ablon G. The Safety and Efficacy of a Proprietary Bioactive Fatty Acids Extract From Saw Palmetto (Serenoa repens) for Promoting Hair Growth and Reducing Hair Loss in Adults With Self-Perceived Thinning Hair: 90-Day Results. J Cosmet Dermatol. 2025 Dec;24(12):e70585. doi: 10.1111/jocd.70585. PMID 41319217